CLINICAL TRIAL: NCT02041702
Title: A Clinical Evaluation of the Safety and Efficacy of St. Jude Medical (SJM) Magnetic Resonance Imaging (MRI) Conditional Pacing System in Patients Undergoing Cardiac MRI
Brief Title: Accent Cardiac MRI Study
Acronym: Accent Cardiac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CR-13-031-AP-LV
Record Dates: First submitted 2013-12-20; First posted 2014-01-22 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Bradycardia
Keywords: Bradycardia; MRI Conditional Pacemaker; St Jude Medical; Accent MRI Pacemaker; Tendril MRI Lead
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cardiac MRI Scan Group (Experimental)
  Interventions: Diagnostic Test: Non-Diagnostic Cardiac MRI scan
- Control Group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Non-Diagnostic Cardiac MRI scan
  Arms: Cardiac MRI Scan Group

SUMMARY:
The aim of this study was to assess safety and efficacy of SJM MRI conditional pacing system. The study hypothesized that cardiac MRI scan would not affect performance of SJM MRI conditional pacing system.

DETAILED DESCRIPTION:
Accent Cardiac MRI study was a prospective, randomized ,multi-center study conducted in Asia. Subjects indicated for dual-chamber pacemaker and who signed study consent form were considered enrolled and post implant were randomized to either Cardiac MRI Scan Group or Control Group.

Clinical evaluation and device interrogation were performed at baseline, pre- and post-MRI scan, and one month post-MRI for all subjects. At 9-12 weeks post-implant, patients in Cardiac MRI Scan Group underwent an elective non-diagnostic cardiac MRI scan at 1.5 Tesla (T) while patients in Control group underwent device interrogation and clinical evaluation twice with a 45-minute waiting period in between. The safety endpoint was freedom from MRI-related complications while efficacy endpoint was change in right atrial/ ventricular (RA/RV) capture threshold and sensing amplitude from pre-MRI scan to one month post-MRI scan.

ELIGIBILITY:
Inclusion Criteria

* Have an approved indication per American College of Cardiology(ACC)/ American Heart Association(AHA)/ Heart Rhythm Society(HRS)/ European Society of Cardiology(ESC) guidelines for implantation of a pacemaker
* Will receive a new dual chamber pacemaker and leads
* Be willing to undergo an elective MRI scan without complete sedation, that is ,under consciousness during MRI scan
* Be able to provide informed consent for study participation
* Be willing and able to comply with the prescribed follow-up tests and schedule of evaluations
* Is not contraindicated for an MRI scan (per the pre-MRI safety screening form)
* Age≥18 years
* Subjects must be able to undergo pectoral implantation

Exclusion Criteria

* Having an existing pacemaker or Implantable Cardioverter Defibrillator (ICD) .A new pacemaker and lead is required for enrollment
* Permanent Atrial Fibrillation/Flutter
* Are medically indicated for an MRI scan at the time of enrollment
* Have an existing active implanted medical device, e.g. neurostimulator, infusion pump etc
* Have a non-MRI compatible device or material implanted
* Have a lead extender or adaptor
* Be unable to fit in MRI bore; will come into contact with the magnet façade inside the MRI bore
* Are currently participating in a clinical investigation that includes an active treatment arm
* Are allergic to dexamethasone sodium phosphate(DSP)
* Are pregnant or planning to become pregnant during the duration of the study
* Have a life expectancy of less than 12 months due to any condition
* Subjects with exclusion criteria required by local law (e.g. age)
* Are unable to comply with the follow up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Keong Ching, Dr, Principal Investigator — National Heart Center Singapore; Rabindra Nath Chakraborty, Dr, Principal Investigator — Apollo Gleneagles Hospital Kolkata India
Locations (13):
- Zhejiang Greentown Cardiovascular Disease Hospital, Hangzhou, China
- Prince of Wales Hospital, Hong Kong, Hong Kong
- India (7):
  - Fortis Hospital, Mohali, Punjab
  - Care Institute of Medical Sciences, Ahmedabad
  - Apollo Hospitals, Bhubaneshwar, Bhubaneshwar
  - Medanta - The Medicity Hospital, Gūrgaon
  - All India Institute of Medical Sciences, New Delhi, New Delhi
  - Fortis Escorts Heart Institute and Research Center, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi
- Serdang Hospital, Kajang, Malaysia
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac MRI Scan Group: Non-diagnostic cardiac MRI scan
- Control Group: No non-diagnostic cardiac MRI scan
Period: Overall Study
Arm/Group | Cardiac MRI Scan Group | Control Group
Started (Enrollment & Baseline) | 140 | 143
Pre MRI Scan/ Pre Waitng (Control Group: No non diagnostic cardiac MRI scan, subjects waited for 45 minutes +/- 15 minutes) | 129 | 140
Post MRI Scan/ Post Waiting (Control Group: No non diagnostic cardiac MRI scan, subjects waited for 45 minutes +/- 15 minutes) | 129 | 140
Completed (One month post MRI Scan) | 129 | 134
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 1 | 6
Not completed — Death | 4 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Patient not confirmed as MRI compatible | 1 | 0
Not completed — Cardiac Resynchronization Therapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac MRI Scan Group | Control Group | Total
Number analyzed (Participants) | 140 | 143 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (11.2) | 67.4 (11.7) | 69.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 82 | 82 | 164
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 15 | 15 | 30
  China | 3 | 4 | 7
  Malaysia | 2 | 3 | 5
  Thailand | 46 | 46 | 92
  India | 54 | 55 | 109
  Singapore | 20 | 20 | 40
Cardiomyopathy History [Count of Participants; unit: Participants]
  Ischemic Cardiomyopathy | 2 | 3 | 5
  Non-ischemic Cardiomyopathy | 1 | 0 | 1
Arrhythmia History [Count of Participants; unit: Participants]
  Atrial Fibrillation | 29 | 26 | 55
  Atrial Flutter | 7 | 6 | 13
  Premature Ventricular | 1 | 2 | 3
  Monomorphic Ventricular Tachycardia | 1 | 0 | 1
  Supraventricular Tachycardia | 1 | 0 | 1
Cardiovascular Medication [Count of Participants; unit: Participants]
  Angiotensin Converting Enzyme Inhibitor | 18 | 17 | 35
  Angiotensin II Receptor Blockers | 31 | 31 | 62
  Beta-Blockers | 31 | 19 | 50
  Aldosterone Inhibitors | 0 | 2 | 2
  Antiarrhythmics (Class I) | 3 | 1 | 4
  Antiarrhythmics (Class II) | 2 | 7 | 9
  Anticoagulants | 15 | 13 | 28
  Antiplatelets | 47 | 48 | 95
  Calcium Channel Blockers | 54 | 40 | 94
  Cardiac Glycosides (Digitalis) | 2 | 1 | 3
  Diuretics | 16 | 16 | 32
  Nitrates | 16 | 9 | 25
  Other Medication | 38 | 29 | 67

OUTCOME MEASURES:

1. Primary Outcome: Freedom From MRI Scan-related Complications
Description: Number of subjects who were free from MRI scan-related complications
Time Frame: MRI Visit ,1 Month Post MRI Visit
Population: All subjects in Cardiac MRI Scan group who underwent an elective non-diagnostic cardiac MRI scan and completed all protocol specific visits were included in the analysis. Subjects who withdrew from the study before 1 month post MRI visit and had no MRI scan related complications were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac MRI Scan Group
Number analyzed (Participants) | 123
Participants | 123
Statistical Analysis 1: Comparison: Cardiac MRI Scan Group; The hypothesis was: H0: P≤ 90% vs H1: P>90% P: The proportion of subjects free from MRI scan related complications at 1 month post MRI scan in cardiac MRI scan group; Test type: Superiority — The 2-sided 90% confidence interval (CI) was calculated using the Clopper-Pearson method; p < 0.01, Clopper-Pearson; Clopper-Pearson CI for the binomial proportion; Ratio = 100, 90% CI 2-sided [97.6 to 100] — The null hypothesis would be rejected if the lower bound of the 2-sided 90% confidence interval was greater than 90%

2. Primary Outcome: Change in Right Atrial (RA) Capture Threshold @0.5 Millisecond (ms) From Pre-MRI Scan to 1 Month After MRI Scan
Description: Number of subjects who experienced an increase in RA capture threshold @ 0.5 ms at 1-Month post MRI scan visit ≤ 0.5 Volt (V) compared to pre-MRI scan value collected at MRI scan visit
Time Frame: MRI Visit ,1 Month Post MRI Visit
Population: Subject successfully implanted, randomized, completed MRI and 1-month post MRI visit, had pre-MRI sensing amplitude ≥ 5 millivolt (mV) in RV &1.5 mV in RA and had an intrinsic rate ≥ 30 beat per minute (bpm) at the time of ventricular sensing amplitude measurement, received an MRI scan if he was in MRI scan group and fulfilled MRI Conditions of Use
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac MRI Scan Group | Control Group
Number analyzed (Participants) | 111 | 117
Participants | 110 | 117
Statistical Analysis 1: Comparison: Cardiac MRI Scan Group vs Control Group; The hypothesis was: H0: PMRI - PCTRL≤ -10% vs H1: PMRI - PCTRL>-10% * PMRI: the success rate in the Cardiac MRI scan group for the change in right atrial capture threshold @0.5ms at 1month post MRI compared to pre-MRI scan value collected at MRI scan visit * PCTRL: the success rate in the Control group for the change in right atrial capture threshold @0.5ms at 1month post MRI compared to pre-MRI scan value collected at MRI scan visit; Test type: Non-Inferiority — The 2-sided 90% CI for difference in success rate between 2 groups was calculated by Farrington-Manning method; p = 0.0007, Farrington-Manning Test; Ratio Difference = -0.9, 90% CI 2-sided [-5.6 to 3.8] — The null hypothesis would be rejected if the lower bound of the two-sided 90% confidence interval was greater than -10%

3. Primary Outcome: Change in Right Ventricular (RV) Capture Threshold @0.5ms From Pre-MRI Scan to 1 Month After MRI Scan
Description: Number of subjects who experienced an increase in RV capture threshold @ 0.5 ms at 1-Month post MRI scan visit ≤ 0.5 V compared to pre-MRI scan value collected at MRI scan visit
Time Frame: MRI Visit, 1 Month Post MRI Visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac MRI Scan Group | Control Group
Number analyzed (Participants) | 120 | 124
Participants | 118 | 124
Statistical Analysis 1: Comparison: Cardiac MRI Scan Group vs Control Group; The hypothesis was: H0: PMRI - PCTRL≤ -10% vs H1: PMRI - PCTRL >-10% * PMRI: the success rate in the Cardiac MRI Scan Group for change in RV capture threshold value @0.5ms at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit * PCTRL: the success rate in Control Group for change in RV capture threshold value @0.5ms at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit; Test type: Non-Inferiority — The 2-sided 90% CI for difference in success rate between 2 groups was calculated by Farrington-Manning method; p = 0.0012, Farrington-Manning test; Ratio Difference = -1.7, 90% CI 2-sided [-6.2 to 2.8] — The null hypothesis would be rejected if the lower bound of the two-sided 90% confidence interval was greater than -10%

4. Primary Outcome: Change in RA Sensing Amplitude From Pre-MRI Scan to 1 Month After MRI Scan
Description: Number of subjects who experienced a decrease in RA sensing amplitude ≤ 50% and at least 1.5 mV at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit
Time Frame: MRI Visit, 1 Month Post MRI Visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac MRI Scan Group | Control Group
Number analyzed (Participants) | 121 | 124
Participants | 105 | 111
Statistical Analysis 1: Comparison: Cardiac MRI Scan Group vs Control Group; The hypothesis was:H0: PMRI - PCTRL≤ -10% vs H1: PMRI - PCTRL >-10% * PMRI: the success rate in MRI Scan Group for change in RA sensing amplitude at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit * PCTRL: the success rate in Control Group for change in RA sensing amplitude at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit; Test type: Non-Inferiority — The 2-sided 90% CI for difference in success rate between 2 groups was calculated by Farrington-Manning method; p = 0.0446, Farrington-Manning test; Ratio Difference = -2.7, 90% CI 2-sided [-9.8 to 4.3] — The null hypothesis would be rejected if the lower bound of the two-sided 90% confidence interval was greater than -10%

5. Primary Outcome: Change in RV Sensing Amplitude From Pre-MRI Scan to 1 Month After MRI Scan
Description: Number of subjects who experienced a decrease in RV sensing amplitude ≤ 50% and at least 5 mV at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit
Time Frame: MRI Visit, 1 Month Post MRI Visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac MRI Scan Group | Control Group
Number analyzed (Participants) | 104 | 111
Participants | 102 | 106
Statistical Analysis 1: Comparison: Cardiac MRI Scan Group vs Control Group; The hypothesis was: H0: PMRI - PCTRL≤ -10% vs H1: PMRI - PCTRL >-10% * PMRI: the success rate in the Cardiac MRI Scan Group for change in RV sensing amplitude at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit * PCTRL: the success rate in the Control Group for change in RV sensing amplitude at 1-Month post MRI scan visit compared to pre-MRI scan value collected at MRI scan visit; Test type: Non-Inferiority — The 2-sided 90% CI for difference in success rate between 2 groups was calculated by Farrington-Manning method; p = 0.0002, Farrington-Manning test; Ratio Difference = 2.6, 90% CI 2-sided [-3.2 to 8.4] — The null hypothesis would be rejected if the lower bound of the two-sided 90% confidence interval was greater than -10%

ADVERSE EVENTS:
Time Frame: Death, Adverse Device Effect (ADE) and Serious Adverse Device Effect (SADE) from Baseline to 1 month post MRI Scan Visit were collected.
Description: 1. In the Serious Adverse Event Section, only SADE are reported.
  2. In the Other (Not Including Serious) Adverse Events Section, only ADE are reported.
  3. In the All-Cause Mortality Section, there are 4 deaths reported. All of them happened prior to cardiac MRI scan and were not related to study procedures.
Arm/Group | Cardiac MRI Scan Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/140 | 0/143
Serious Adverse Events (participants affected / at risk) | 6/140 | 6/143
Other Adverse Events (participants affected / at risk) | 1/140 | 1/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac MRI Scan Group (N=140) | Control Group (N=143)
Acute Non-St Elevation Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anaphylaxis, Anaphylactoid (General disorders) | 1 (1) | 0 (0)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dressler's Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Drug Allergy (General disorders) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Righ Atrial Lead Dislodgement (Cardiac disorders) | 0 (0) | 2 (2)
Right Ventricular Lead Dislodgement (Cardiac disorders) | 1 (1) | 0 (0)
System Infection (Infections and infestations) | 0 (0) | 1 (1)
Ventricular Tachycardia Requiring Emergent Direct Current Cardioversion (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardiac MRI Scan Group (N=140) | Control Group (N=143)
New Onset Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Retracted Right Atrial Lead (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less